CLINICAL TRIAL: NCT00360360
Title: A Phase II Study of Paclitaxel/Carboplatin Plus Bevacizumab/Erlotinib in the First Line Treatment of Patients With Carcinoma of Unknown Primary Site
Brief Title: Paclitaxel/Carboplatin Plus Bevacizumab/Erlotinib in the First Line Treatment of Carcinoma of Unknown Primary Site
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI UNKPRI 19
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Neoplasm, Unknown Primary
Keywords: Neoplasm, Unknown Primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Paclitaxel; Carboplatin; Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab/Paclitaxel/Carboplatin/Erlotinib (Experimental): Bevacizumab 15mg/kg IV infusion,Day 1 Paclitaxel 175mg/m2, 1-3 hour IV infusion,Day 1 Carboplatin AUC 6.0 IV Day 1 Erlotinib 150 mg by mouth daily
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: bevacizumab; Drug: erlotinib

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel 175mg/m2, 1-3 hour IV infusion,Day 1
  Other Names: Taxol
Drug: carboplatin — Carboplatin AUC 6.0 IV Day 1
  Other Names: Paraplatin
Drug: bevacizumab — Bevacizumab 15mg/kg IV infusion,Day 1
  Other Names: Avastin
Drug: erlotinib — Erlotinib 150 mg by mouth daily
  Other Names: Tarceva

SUMMARY:
We will evaluate the feasibility, toxicity, and effectiveness of combination chemotherapy (paclitaxel/carboplatin)plus combination targeted therapy (bevacizumab/erlotinib)in the first line treatment of patients with carcinoma of unknown primary site. There is limited experience with either bevacizumab or erlotinib in the treatment of cancers of unknown site but given the heterogeneous nature of the tumor, it is likely that inhibition of angiogenesis pathways and/or the EGFR pathway are effective strategies in at least a proportion.

DETAILED DESCRIPTION:
All eligible patients will receive:

* Bevacizumab 15mg/kg IV infusion,Day 1
* Paclitaxel 175mg/m2, 1-3 hour IV infusion,Day 1
* Carboplatin AUC 6.0 IV Day 1
* Erlotinib 150 mg by mouth daily

The regimen will be repeated every 21 days for a total of 4 courses. Patients will be initially evaluated for response after completing 2 courses (6 weeks) of treatment. Patients with an objective tumor response or stable disease will continue treatment for another 2 courses. Patients will be re-evaluated after 4 courses and those with objective tumor response or stable disease will stop chemotherapy with paclitaxel/carboplatin and continue treatment with bevacizumab/erlotinib until tumor progression is documented for a maximum of 12 months. During treatment with bevacizumab/erlotinib response will be evaluated every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven metastatic carcinoma with the following light microscopic histologies: adenocarcinoma, poorly differentiated carcinoma(must have immunoperoxidase stains to rule out lymphoma, neuroendocrine carcinoma),or poorly differentiated squamous carcinoma.
* ECOG performance status 0-1
* No previous treatment with any systemic therapy
* Adequate kidney, liver and bone marrow function
* Be able to understand the nature of the study and give written informed consent

Exclusion Criteria:

* The following specific syndromes:
* Neuroendocrine carcinoma
* Women with adenocarcinoma isolated to axillary lymph nodes
* Women with adenocarcinoma isolated to peritoneal involvement
* Carcinoma involving only one site with resectable tumors at that site
* Squamous carcinoma limited to cervical, supraclavicular, or inguinal lymph nodes
* Uncontrolled brain metastases and all patients with meningeal involvement
* Women pregnant or lactating
* Clinically significant cardiovascular disease
* History of myocardial infarction or stroke within 6 months
* Clinical history of hemoptysis or hematemesis
* Patients with PEG tubes or G-tubes
* Proteinuria
* History of bleeding diathesis or coagulopathy

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-07; Primary Completion 2008-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (9):
- United States (9):
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Hainsworth JD, Spigel DR, Thompson DS, Murphy PB, Lane CM, Waterhouse DM, Naot Y, Greco FA. Paclitaxel/carboplatin plus bevacizumab/erlotinib in the first-line treatment of patients with carcinoma of unknown primary site. Oncologist. 2009 Dec;14(12):1189-97. doi: 10.1634/theoncologist.2009-0112. Epub 2009 Dec 4. PMID 19965914

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab/Paclitaxel/Carboplatin/Erlotinib
Started | 60
Completed | 54
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab/Paclitaxel/Carboplatin/Erlotinib
Number analyzed (Participants) | 60
Age Continuous [Median (Full Range); unit: years] | 50 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Paclitaxel/Carboplatin/Erlotinib
Number analyzed (Participants) | 54
months | 12.6 [9.7 to 18.5]

2. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab/Paclitaxel/Carboplatin/Erlotinib
Number analyzed (Participants) | 54
months | 8 [6.4 to 13.8]

ADVERSE EVENTS:
Arm/Group | Bevacizumab/Paclitaxel/Carboplatin/Erlotinib
Serious Adverse Events (participants affected / at risk) | 29/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Paclitaxel/Carboplatin/Erlotinib (N=60)
Acidosis (Metabolism and nutrition disorders) | 1 (1) — Diabetic ketoacidosis
Dehydration (Gastrointestinal disorders) | 7 (11)
Febrile neutropenia (Infections and infestations) | 5 (5)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Neuroendocrine: ADH secretion abnormality (Endocrine disorders) | 1 (1) — SIADH
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Anterior chest discomfort
Cardiac General (Cardiac disorders) | 1 (1) — Cardiogenic shock
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — Cellulitis
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) — Orthostatic
Perforation (Gastrointestinal disorders) | 1 (1) — Sigmoid perforation
Pain (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (3)
Obstruction, GI (Gastrointestinal disorders) | 1 (1) — Small bowel obstruction
Pericardial tumor constriction (Cardiac disorders) | 1 (1)
Pain (Gastrointestinal disorders) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia
Hemorrhage (Gastrointestinal disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) — Bradycardia
CNS cerebrovascular ischemia (Vascular disorders) | 1 (1) — TIA
Generalized weakness (General disorders) | 1 (1)
disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab/Paclitaxel/Carboplatin/Erlotinib (N=60)
Rash (acneiform) (Skin and subcutaneous tissue disorders) | 5 (7)
Allergic Reaction/Hypersensitivity Grade (Immune system disorders) | 6 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 27 (94)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Anorexia (Gastrointestinal disorders) | 31 (90)
Bleeding (gums) (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 23 (45)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (20)
Dehydration (Gastrointestinal disorders) | 16 (34)
Depression (Psychiatric disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 40 (139)
Dizziness/Lightheadedness (Nervous system disorders) | 5 (10)
Dyspepsia (Gastrointestinal disorders) | 3 (8)
Dysphagia (Gastrointestinal disorders) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (42)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 (28)
Fatigue (General disorders) | 45 (237)
Fever (General disorders) | 8 (8)
Headache (Nervous system disorders) | 12 (31)
Hemoglobin (Metabolism and nutrition disorders) | 34 (124)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (16)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (12)
Hypertension (Cardiac disorders) | 4 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Hypotension (Cardiac disorders) | 17 (55)
Indigestion (Gastrointestinal disorders) | 3 (15)
Insomnia (General disorders) | 9 (24)
Leukocytes (WBC) (Blood and lymphatic system disorders) | 28 (61)
Mood alteration (anxiety) (Psychiatric disorders) | 7 (15)
Mood alteration (confusion) (Psychiatric disorders) | 3 (4)
Mood alteration (depression) (Psychiatric disorders) | 5 (6)
Mouth (sore) (Gastrointestinal disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 8 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (34)
Nausea (Gastrointestinal disorders) | 40 (125)
Neuropathy-sensory (Nervous system disorders) | 19 (101)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenic fever (Infections and infestations) | 3 (3)
Neutrophils (ANC) (Blood and lymphatic system disorders) | 30 (53)
Night Sweats (General disorders) | 3 (3)
Pain (NOS) (General disorders) | 3 (5)
Pain (abdominal) (Gastrointestinal disorders) | 10 (15)
Pain (back) (Musculoskeletal and connective tissue disorders) | 5 (20)
Pain (bone) (Musculoskeletal and connective tissue disorders) | 6 (8)
Pain (chest) (Cardiac disorders) | 3 (3)
Pain (legs) (Musculoskeletal and connective tissue disorders) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 31 (77)
Proteinuria (Metabolism and nutrition disorders) | 12 (20)
Pruritis (Skin and subcutaneous tissue disorders) | 16 (27)
Rash (facial) (Skin and subcutaneous tissue disorders) | 3 (5)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 45 (218)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Skin (dry) (Skin and subcutaneous tissue disorders) | 7 (20)
Taste alteration (Gastrointestinal disorders) | 6 (14)
Throat (sore) (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Weight Loss (General disorders) | 9 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.